CLINICAL TRIAL: NCT07344753
Title: 20 000 Lieues Sous l'IRM - New Simulation Care Pathway for Paediatric MRI Preparation : Exploratory Descriptive Pilot Study
Brief Title: New Simulation Care Pathway for Paediatric MRI Preparation
Status: Not yet recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: Direction Générale de l'offre de Soins (DGOS) (Unknown)
Responsible Party: Sponsor
Other Study IDs: RC25_0371
Record Dates: First submitted 2026-01-07; First posted 2026-01-15 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Magnetic Resonance Imaging (MRI)
Keywords: Magnetic Resonance Imaging (MRI); Immersive experience; Paediatric MRI

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study patient
  Interventions: Other: Realization of the immersive experience; Other: Completion of study questionnaires; Other: Questioning the child's emotional feelings

INTERVENTIONS:
Other: Realization of the immersive experience — The immersive experience is divided into four modules, to be completed in the following order:
  First module: the tunnel (confinement) The child lies down on the mat, and the paramedical staff slowly slide the tunnel over them until their head is in the middle of it.
  Second module: noise. The child must press three illuminated buttons that produce the sounds of an MRI scan (recorded by us).
  Third module: the diving suit (equipment constraints) In order to use the submarine, the child must wear noise-cancelling headphones. They stand against the wall and the professional helps them to put the headphones on correctly over their ears.
  Fourth module: static position (immobility). The child lies down on a mat in a mould that fits their size (3 sizes available). They watch an animated film lasting 3 minutes 30 seconds (the average duration of an MRI sequence). Their body must not move out of the mould, proving that they have managed to remain still.
Other: Completion of study questionnaires — Assessment of the child's satisfaction with each module using a simplified 3-point scale adapted to very young children (positive, neutral, negative experience) Assessment of the guardian's satisfaction through a series of questions following the immersive experience and the MRI scan
Other: Questioning the child's emotional feelings — The child's emotional response, recorded using an emotion weather chart (4 icons) before and after the immersive experience and before and after the MRI scan.

SUMMARY:
Magnetic resonance imaging (MRI) is a common imaging procedure that is safe and non-invasive, as it relies on the use of different magnetic fields. It is the gold standard examination for a wide range of pathologies.

However, it has many disadvantages, including the repetitive noise produced by the coils during image acquisition sequences, which can cause discomfort. The noise level often exceeds 100 dB, while the noise exposure limit for workers is set at 87 dB. There is no regulatory limit for patients. Although it is relatively loud and quite unpleasant, this noise is not harmful to health and does not amplify, contrary to the perception that one may have in the tunnel. Noise-cancelling headphones and earbuds are strongly recommended for patients to reduce any discomfort that may result. In practice, the imaging department requires all patients to wear hearing protection.

Other disadvantages of MRI include confinement in a tunnel and the need to remain completely immobile for approximately six sequences, each of 2 to 5 minutes in duration.

This can be problematic, particularly for patients suffering from pain or respiratory failure, or for agitated individuals who find it difficult to remain motionless in a lying position for long periods of time.

These various issues are particularly relevant in the paediatric population, for whom MRI is the preferred imaging technique due to its safety in terms of radiation exposure.

The specific characteristics of this population require more complex patient management due to the particular constraints of MRI. Acceptance of the following four points appears to be key to its successful implementation: lying down, with the head in a tunnel, intense and repeated noises, and strict immobility for at least 30 minutes. Without these conditions, the images recorded will not provide reliable results that can be used for diagnosis.

To meet these constraints, at Nantes University Hospital, general anaesthesia was routinely administered to children aged 3 to 6 until September 2023. This ensures a 100% success rate for the examination, but it is not a trivial procedure for the child and is stressful for their parents. Since then, a light sedation protocol has been offered as part of the care pathway. This involves the child taking medication one hour and then thirty minutes before the MRI scan to calm them down until they fall asleep.

Unfortunately, access to this MRI under light sedation or general anaesthesia complicates the appointment booking process, as it requires the presence of a medical team during dedicated shifts.

MRI scans under light sedation are scheduled for three slots per week. At the end of 2025, the waiting time was four months for light sedation and six months for general anaesthesia.

In order to improve and speed up the care of children who need to perform an MRI scan, a specific consultation with an immersive four-module programme has been designed at Nantes University Hospital with the aim of optimising the chances of success of the examination without general anaesthesia or sedation, thereby:

* Reduce waiting times for appointments, and thus reduce the period of stress for parents awaiting a diagnosis for their child.
* Reduce the time required for the examination. Indeed, an examination under light sedation considerably lengthens the treatment time, with a sedation onset time of approximately 1.5 hours.
* Increasing the success rate of MRI scans under light sedation following failure without sedation.

This innovative approach is based on an immersive experience in the form of a course consisting of four modules designed to help children practise four areas that can be challenging for them (immersion in a tunnel, loud noise, the constraints of specific equipment, and immobility). These modules are themed around the marine world, in line with the already approved paediatric radiology programme. It will be offered to children aged 3 to 6 with no cognitive or behavioural disorders.

The modules will be installed in a paediatric consultation room and will be used for half a day each month. When not needed, they'll be put away so the room can be used for consultations.

The aim of our pilot study is to assess the impact of this immersive journey on the success of an MRI scan without general anaesthesia or sedation.

ELIGIBILITY:
Inclusion criteria

* Children aged 36 to 72 months scheduled to undergo an MRI scan
* Consent obtained from the child and their parent or legal guardian
* Patient affiliated with the social security system, CMU
* Children undergoing an MRI scan for the first time Exclusion criteria
* Children who are completely hostile to the experience.
* Children with cognitive or behavioural disorders.
* Children or parents/guardians who do not understand French.
* Children coming to validate the fitting of a cochlear implant

Ages: 36 Months to 72 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study will focus on children aged between 3 and 6 years old who are scheduled to undergo an MRI scan (any anatomical region).
Sampling Method: Probability Sample
Enrollment: 114 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2028-08-15 (Estimated); Study Completion 2028-08-15 (Estimated)

PRIMARY OUTCOMES:
Assess the usefulness of an immersive experience in the success of an MRI scan on the first attempt without general anaesthesia or sedation for children aged 3 to 6 years. | 14 days
  Our main criteria is obtaining a diagnosis (pathological or otherwise) following an MRI scan using the immersive approach. Children who have not completed the immersive approach and therefore have not undergone an MRI scan without general anaesthesia or sedation will be considered to have been unsuccessful. In addition, children who have successfully completed the immersive pathway but whose MRI scan without general anaesthesia or sedation does not result in a diagnosis (and for whom an additional MRI scan must therefore be scheduled) will be considered unsuccessful.

SECONDARY OUTCOMES:
Assess the success rate of MRI without general anaesthesia or sedation in the subgroup of children who successfully completed the immersive experience. | 14 days
Description of the implementation of the four modules of the immersive experience (proportion of patients who failed each module) | 14 days
Assessment of the patient's emotional response to the immersive experience and the MRI scan with an emotional weather forecast (4 icons) before and after the immersive experience, as well as before and after the MRI scan | 14 days
Assess patient satisfaction with the immersive experience based on a simplified 3-point facial expression scale adapted to very young children (positive, neutral, negative experiences) | 1 day
Research of factors associated with successful MRI without general anaesthesia or sedation. | 14 days
  The success of the MRI is defined in the main criteria. The factors studied to predict this will be: success or failure in each module of the immersion programme, the number of modules completed, the child's age, gender, schooling, childcare arrangements prior to schooling, and the positive or negative assessment of the immersion programme by the child and parents.
Assessment of tutors' satisfaction with the immersive programme and the performance of MRI. | 14 days
Assessment of the hospital cost of the immersive procedure and MRI depending on the conditions (with/without general anaesthesia or sedation): professional time, cost of immersive modules, drugs/devices for anaesthesia/sedation and monitoring. | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Ribbe, Principal Investigator — Nantes University Hospital; Lucie Breteau, Principal Investigator — Nantes University Hospital; Stéphanie Hatron, Principal Investigator — Nantes University Hospital

IPD SHARING:
Plan to Share IPD: Undecided